CLINICAL TRIAL: NCT05861011
Title: Surgical Outcomes of Bladder Neck Procedures in Children With Neurogenic Bladder: a Retrospective Monocentric Study
Brief Title: Bladder Neck Surgery in Children With Neurogenic Bladder
Acronym: CERPED
Status: Completed | Type: Observational
Sponsor: University of Lorraine (Other)
Responsible Party: Principal Investigator, Dr Christelle DESTINVAL, Principal Investigator, University of Lorraine
Other Study IDs: ULora; 2023PI004 (Registry Identifier: DRCI)
Record Dates: First submitted 2023-04-13; First posted 2023-05-16 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Incontinence, Urinary; Bladder Dysfunction; Spina Bifida; Neurogenic Bladder
Keywords: Bladder Neck Surgery; Children; Surgical Outcomes; Retrospective Study
MeSH Terms: conditions — Urinary Incontinence; Spinal Dysraphism; Urinary Bladder, Neurogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Surgical outcomes of bladder neck surgery in children with neurogenic bladder.

Consequences on bladder voiding.

DETAILED DESCRIPTION:
Surgical outcomes of bladder neck surgery in children with neurogenic bladder:

Quality of voiding: spontaneous, need for catheterization, or incontinence.

Other surgical complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients, with neurogenic bladder and younger than 18 years old ,who underwent a bladder neck procedure

Exclusion Criteria:

* Patients, with neurogenic bladder and older than 18 years old ,who underwent a bladder neck procedure

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients with neurogenic bladder
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Number of participants with delayed or incomplete opening of the bladder neck during the voiding phase of micturition impeding urine flow | Baseline (Before surgery)
  Cysto-urethrogram and uroflowmetry help diagnose delayed or incomplete opening of the bladder neck.
  delayed or incomplete opening of the bladder neck
Number of participants with muscular bladder | Baseline (Before surgery)
  The muscular bladder has thicker walls, bladder diverticula and trabecules (diagnosed during abdominal ultrasound, urethro-cystogram and cystoscopy)

SECONDARY OUTCOMES:
Length of stay | From admission to discharge home, up to 20 days
  Length of stay
The time length between the surgery date and the postoperative consultation date | Through study completion, an average of 2 years
  Follow_up represents the time length between the surgery date and the postoperative consultation date in days, months, or years. Generally, there are a-month-follow-up, a three month-follow-up, a six month-follow-up, and a year-follow-up. The surgeon can see the patient if there is any problem between these consultations. After a year of follow-up, it is up to the surgeon to decide if the patient needs to be seen yearly or not. The last follow-up date is crucial because it indicates how the patient is and if other follow-up dates need to be applied.
Surgical complications after bladder neck procedure | Through study completion, an average of 2 years
  bleeding, bowel obstruction, surgical hernia, urinary stone, urinary infection
Operating time | Intraoperative
  Operating time

CONTACTS AND LOCATIONS:
Overall Officials: Christelle Destinval, MD, Principal Investigator — University of Lorraine
Locations (1):
- ULorraine, Vandœuvre-lès-Nancy, Grand Est, France

IPD SHARING:
Plan to Share IPD: No
In the name of anonymization, the investigators won't share individual participant data

REFERENCES:
- [Background] Stein R, Bogaert G, Dogan HS, Hoen L, Kocvara R, Nijman RJM, Quaedackers J, Rawashdeh YF, Silay MS, Tekgul S, Radmayr C. EAU/ESPU guidelines on the management of neurogenic bladder in children and adolescent part II operative management. Neurourol Urodyn. 2020 Feb;39(2):498-506. doi: 10.1002/nau.24248. Epub 2019 Dec 3. PMID 31794087